CLINICAL TRIAL: NCT00699491
Title: Phase I/II Trial of IMC-A12 in Combination With Temsirolimus in Patients With Metastatic Breast Cancer
Brief Title: Cixutumumab and Temsirolimus in Treating Patients With Locally Recurrent or Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00284; NCI-2009-00284 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000598057; MC0736 (Other: Alliance for Clinical Trials in Oncology); 8129 (Other: CTEP); N01CM00071 (NIH); N01CM00099 (NIH); N01CM62201 (NIH); N01CM62205 (NIH); N01CM62207 (NIH); N01CM62209 (NIH); U10CA180821 (NIH); U10CA025224 (NIH)
Record Dates: First submitted 2008-06-17; First posted 2008-06-18 (Estimated); Results first posted 2015-05-21 (Estimated); Last update posted 2018-06-13 (Actual); Status verified 2018-05

CONDITIONS: Male Breast Carcinoma; Recurrent Breast Carcinoma; Stage IV Breast Cancer AJCC v6 and v7
MeSH Terms: conditions — Breast Neoplasms, Male; Breast Neoplasms | interventions — cixutumumab; temsirolimus; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (cixutumumab, temsirolimus) (Experimental): Patients receive temsirolimus IV over 30 minutes and cixutumumab IV over 60 minutes on days 1, 8, 15, and 22 (cixutumumab is given on days 8, 15, and 22 of course 1 only). Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Cixutumumab; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Temsirolimus

INTERVENTIONS:
Biological: Cixutumumab — Given IV
  Other Names: Anti-IGF-1R Recombinant Monoclonal Antibody IMC-A12; IMC-A12
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Drug: Temsirolimus — Given IV
  Other Names: CCI-779; CCI-779 Rapamycin Analog; Cell Cycle Inhibitor 779; Rapamycin Analog; Rapamycin Analog CCI-779; Torisel

SUMMARY:
This phase I/II trial is studying the side effects and best dose of cixutumumab when given together with temsirolimus and to see how well they work in treating patients with breast cancer that has recurred (come back) at or near the same place as the original (primary) tumor or has spread to other places in the body. Monoclonal antibodies, such as cixutumumab, can block tumor growth in different ways by targeting certain cells. Temsirolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving cixutumumab together with temsirolimus may be a better treatment for breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To establish the recommended dose level for the phase II trial. (Phase I) II. To examine the safety profile of this combination in patients with metastatic breast cancer. (Phase I) III. To assess the anti-tumor activity (in terms of overall response rate) and toxicity profile of IMC-A12 (cixutumumab) in combination with temsirolimus in patients with metastatic breast cancer. (Phase II)

SECONDARY OBJECTIVES:

I. To estimate the progression-free survival (PFS) and overall survival distributions (as well as the 6-month PFS rate).

II. To evaluate the in vivo mechanisms of action of temsirolimus in combination with IMC-A12 and to examine potential biomarker predictors of treatment response.

OUTLINE: This is a phase I, dose-escalation study of cixutumumab followed by a phase II study.

Patients receive temsirolimus intravenously (IV) over 30 minutes and cixutumumab IV over 60 minutes on days 1, 8, 15, and 22 (cixutumumab is given on days 8, 15, and 22 of course 1 only). Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically for up to 2 (phase I) or 5 (phase II) years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of breast cancer with diagnosis of metastatic or locally recurrent disease (locally recurrent disease should be stage IV e.g. chest wall involvement)
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1 (Karnofsky >= 80%)
* Life expectancy of > 12 weeks
* Capable of understanding investigational nature, potential risks and benefits of the study and able to provide written informed consent
* Negative serum pregnancy test =< 7 days of registration for women of childbearing potential:

  * Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) for the duration of study therapy and for 3 months after the last dose of IMC-A12 and CCI-779 (temsirolimus)
  * Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
  * Nursing women must be willing to discontinue nursing; NOTE: breastfeeding should be discontinued if the mother is treated with CCI-779 and IMC-A12
* Absolute neutrophil count >= 1,500/mcL
* Hemoglobin >= 8.5 g/dL
* Platelets >= 100,000/mcL
* Total bilirubin =< 1.5 X institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT)(serum glutamate pyruvate transaminase [SGPT]) =< 3 x institutional ULN (=< 5 X institutional ULN if liver function test [LFT] elevations due to liver metastases)
* Creatinine =< 1.5 X institutional ULN OR creatinine clearance >= 60 mL/min/1.73^2 for patients with creatinine > institutional ULN
* Fasting serum cholesterol =< 350 mg/dL (9.0 mmol/L)
* Fasting triglycerides =< 400 mg/dL (4.56 mmol/L)
* Albumin >= 3.4 mg/dL
* Fasting or non fasting serum glucose < 120 mg/dL
* Hemoglobin A1c (HbA1c) (for all patients with a history of diabetes mellitus) < 8%
* Phase I only: Any number of prior therapy regimens is allowed
* Phase II only: Measurable disease is required for the Phase II portion of the study; measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 20 mm with conventional techniques (computed tomography [CT], magnetic resonance imaging [MRI], x-ray) or as >= 10 mm with spiral CT scan
* Phase II only: =< two and at least one prior chemotherapy regimens in the setting of metastatic or locally recurrent (stage IV chest wall involvement) disease are required

Exclusion Criteria:

* Phase I patients only: Patients with base line diabetes requiring oral hypoglycemics or insulin
* Phase II patients only: Poorly controlled diabetes mellitus; NOTE: patients with a history of diabetes mellitus on oral hypoglycemics or insulin are allowed to participate, provided that their fasting blood glucose is < 120 mg/dL and that they are on a stable dietary or therapeutic regimen for this condition
* Any of the following:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception (hormonal agents are not allowed and oral contraceptives are not acceptable for contraception)
* Receiving hormonal agents used for the treatment of breast cancer with the exception that premenopausal women who have been on a gonadotropin-releasing hormone (GnRH) agonist and subsequently progressed may, at the discretion of the treating physician, continue on the GnRH agonist
* Any of the following prior therapies:

  * Systemic anti-cancer therapy =< 3 weeks prior to registration
  * Radiation therapy =< 2 weeks prior to registration
* Prior invasive non-breast malignancy, except for adequately treated basal or squamous cell carcinoma of the skin or other cancer from which the patient has been disease free for >= 5 years
* Known hypersensitivity reactions to macrolide antibiotics (such as erythromycin, clarithromycin, and azithromycin); allergic reactions attributed to compounds of similar chemical or biologic composition to IMC-A12, or temsirolimus
* Prior treatment with agents targeting the insulin-like growth factor-I receptor (IGF-IR)/insulin-like growth factors (IGFs) or phosphatidylinositol-4,5-bisphosphate 3-kinase, catalytic subunit alpha (PI3K)/v-akt murine thymoma viral oncogene homolog 1 (Akt)/mechanistic target of rapamycin (mTOR) pathway
* Receiving any other investigational agents or herbal preparations
* Patients may not be taking oral corticosteroids except for replacement for adrenal insufficiency
* Uncontrolled brain metastases; Note: brain metastases are not permitted on study unless the metastases have been treated by surgery or radiotherapy, and the patient has been neurologically stable and off of steroids for >= 12 weeks
* Known human immunodeficiency virus (HIV)-positive patients who have cluster of differentiation (CD)4 counts below the normal range or who are on anti-retroviral therapy that may interfere with the metabolism of temsirolimus
* Uncontrolled intercurrent illness including, but not limited to:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Uncontrolled symptomatic cardiac arrhythmia
  * Psychiatric illness/social situations that would limit compliance with study requirements
* Receiving enzyme-inducing antiepileptic drugs (EIAEDs; e.g., phenytoin, carbamazepine, phenobarbital) or any other cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4) inducer such as rifampin or St. John's wort

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2008-10-31 (Actual); Primary Completion 2013-09-09 (Actual); Study Completion 2018-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Ma, Principal Investigator — Alliance for Clinical Trials in Oncology
Locations (192):
- United States (192):
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Valley Medical Oncology Consultants, Pleasanton, California
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - SCL Health Saint Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Colorado Cancer Research Program NCORP, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - SCL Health Lutheran Medical Center, Wheat Ridge, Colorado
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Florida Hospital Orlando, Orlando, Florida
  - John B Amos Cancer Center, Columbus, Georgia
  - Hawaii Cancer Care Inc-POB II, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Oncology Inc-Kuakini, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Castle Medical Center, Kailua, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Hawaii Oncology Inc-Pali Momi, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Rush - Copley Medical Center, Aurora, Illinois
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Graham Hospital Association, Canton, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Memorial Hospital, Carthage, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Weiss Memorial Hospital, Chicago, Illinois
  - Heartland Cancer Research NCORP, Decatur, Illinois
  - Eureka Hospital, Eureka, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Illinois CancerCare-Havana, Havana, Illinois
  - Mason District Hospital, Havana, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Mcdonough District Hospital, Macomb, Illinois
  - Holy Family Medical Center, Monmouth, Illinois
  - Illinois CancerCare-Monmouth, Monmouth, Illinois
  - Bromenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center Foundation, Normal, Illinois
  - Illinois CancerCare-Community Cancer Center, Normal, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin Cancer Treatment Center, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois Valley Hospital, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Illinois CancerCare-Spring Valley, Spring Valley, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - Reid Health, Richmond, Indiana
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Kansas City NCI Community Oncology Research Program, Prairie Village, Kansas
  - Union Hospital of Cecil County, Elkton, Maryland
  - Bixby Medical Center, Adrian, Michigan
  - Hickman Cancer Center, Adrian, Michigan
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Beaumont Hospital-Dearborn, Dearborn, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Green Bay Oncology - Escanaba, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center-West Flint Campus, Flint, Michigan
  - Green Bay Oncology - Iron Mountain, Iron Mountain, Michigan
  - Allegiance Health, Jackson, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Mercy Memorial Hospital, Monroe, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Saint Cloud Hospital, Saint Cloud, Minnesota
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Heartland Hematology and Oncology Associates Incorporated, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Saint Joseph Oncology Inc, Saint Joseph, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Nebraska Cancer Research Center, Lincoln, Nebraska
  - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Glens Falls Hospital, Glens Falls, New York
  - Randolph Hospital, Asheboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Annie Penn Memorial Hospital, Reidsville, North Carolina
  - Mid Dakota Clinic, Bismarck, North Dakota
  - Saint Alexius Medical Center, Bismarck, North Dakota
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Altru Cancer Center, Grand Forks, North Dakota
  - Toledo Clinic Cancer Centers-Bowling Green, Bowling Green, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus NCI Community Oncology Research Program, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Health Center, Dayton, Ohio
  - Dayton NCI Community Oncology Research Program, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Hematology Oncology Center Incorporated, Elyria, Ohio
  - Mercy Cancer Center-Elyria, Elyria, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Toledo Clinic Cancer Centers-Oregon, Oregon, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Flower Hospital, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - The Toledo Hospital/Toledo Children's Hospital, Toledo, Ohio
  - Saint Vincent Mercy Medical Center, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - Toledo Community Hospital Oncology Program CCOP, Toledo, Ohio
  - Mercy Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Greene Memorial Hospital, Xenia, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Natalie Warren Bryant Cancer Center at Saint Francis, Tulsa, Oklahoma
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Fredericksburg Oncology Inc, Fredericksburg, Virginia
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Green Bay Oncology - Oconto Falls, Oconto Falls, Wisconsin
  - HSHS Saint Nicholas Hospital, Sheboygan, Wisconsin
  - Green Bay Oncology - Sturgeon Bay, Sturgeon Bay, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level 1: * 25 mg temsirolimus IV over 30 minutes on days 1, 8, 15, and 22
  * 3 mg/ks cixutumumab IV over 60 minutes on days 1, 8, 15, and 22
  Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
- Dose Level -1: * 20 mg temsirolimus IV over 30 minutes on days 1, 8, 15, and 22
  * 3 mg/ks cixutumumab IV over 60 minutes on days 1, 8, 15, and 22
  Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
- Dose Level -2: * 15 mg temsirolimus IV over 30 minutes on days 1, 8, 15, and 22
  * 3 mg/ks cixutumumab IV over 60 minutes on days 1, 8, 15, and 22
  Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
- Dose Level -2A: * 15 mg temsirolimus IV over 30 minutes on days 1, 8, 15, and 22
  * 4 mg/ks cixutumumab IV over 60 minutes on days 1, 8, 15, and 22
  Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
- Dose Level -2B: * 15 mg temsirolimus IV over 30 minutes on days 1, 8, 15, and 22
  * 5 mg/ks cixutumumab IV over 60 minutes on days 1, 8, 15, and 22
  Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
- Phase II: Phase II patients receive the recommended phase II dose determined in the phase I portion.
  * 15 mg temsirolimus IV over 30 minutes on days 1, 8, 15, and 22.
  * 4 mg/kg cixutumumab IV over 60 minutes on days 1, 8, 15, and 22.
  Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Dose Level 1 | Dose Level -1 | Dose Level -2 | Dose Level -2A | Dose Level -2B | Phase II
Started | 3 | 2 | 7 | 6 | 8 | 22
Completed | 3 | 2 | 7 | 6 | 8 | 22
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Level 1 | Dose Level -1 | Dose Level -2 | Dose Level -2A | Dose Level -2B | Phase II | Total
Number analyzed (Participants) | 3 | 2 | 7 | 6 | 8 | 22 | 48
Age, Continuous [Median (Full Range); unit: years] | 35 [34 to 40] | 68 [56 to 80] | 49 [36 to 65] | 53 [43 to 63] | 48.5 [35 to 72] | 57 [35 to 82] | 48.5 [34 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 7 | 6 | 8 | 22 | 48
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 2 | 7 | 6 | 8 | 22 | 48

OUTCOME MEASURES:

1. Primary Outcome: Recommended Dose Level for Phase II Testing (RPTD) (Phase I)
Description: The RPTD is defined as the highest dose level at which at most one of 6 patients develops a dose limiting toxicity (DLT) during the first course of treatment and the next highest dose level has 2 or more DLTs. The number of patients in each cohort reporting a DLT is reported.
  Dose-limiting toxicities (DLTs) are defined as any of the following adverse events (AEs) that are related to study agent with an attribution of possible, probably, or definite and fulfilling one of the following criteria:
  * Any grade 4 hematologic toxicity
  * Hyperglycemia that cannot be stably controlled with diabetic medication
  * Any grade 3 or 4 non-hematologic toxicity (except asymptomatic medically manageable laboratory abnormalities such as hyperlipidemia, hypophosphatemia, and hypokalemia)
Time Frame: During first course
Population: Patients registered to the Phase I portion of the protocol were analyzed for this endpoint. One patient in Dose Level -1, one patient in Dose Level -2, and two patients in Dose Level -2B discontinued study treatment during Cycle 1 for reasons unrelated to toxicity and were excluded from this endpoint.
Measure: Number; unit: DLTs
Arm/Group | Dose Level 1 | Dose Level -1 | Dose Level -2 | Dose Level -2A | Dose Level -2B
Number analyzed (Participants) | 3 | 1 | 6 | 6 | 6
DLTs | 2 | 1 | 1 | 0 | 3

2. Primary Outcome: Tumor Response Rate (TRR) (Complete Response [CR] or Partial Response [PR]) by the Response Evaluation Criteria in Solid Tumors (RECIST) (Phase II)
Description: A response is defined as a disease burden that meets the RECIST criteria for Complete Response (CR) or Partial Response (PR) on 2 consecutive evaluations at least 6-8 weeks apart.
  Complete Response (CR): All of the following must be true:
  1. Disappearance of all target and non-target lesions.
  2. Each target lymph node must have reduction in short axis to <1.0 cm.
  Partial Response (PR): At least a 30% decrease in PBSD (sum of the longest diameter for all target lesions plus the sum of the short axis of all the target lymph nodes at current evaluation) taking as reference the baseline measures.
  The rate is calculated by dividing the number of patients with a CR or PR by the number of evaluable patients. A ninety percent confidence interval for the true tumor response rate will be calculated using the Duffy-Santer approach.
Time Frame: Up to 5 years
Population: One patient registered to the Phase II portion of the study was not eligible for this endpoint due to eligibility criteria not being met.
Measure: Number (90% Confidence Interval); unit: percentage of patients with response
Arm/Group | Phase II
Number analyzed (Participants) | 21
percentage of patients with response | 0 [0 to 13.3]

3. Secondary Outcome: Adverse Events Graded Using the NCI CTCAE Version. 3 (Phase II)
Description: Adverse events will be graded using the NCI-CTCAE v3.0 coding scheme. The maximum grade for each adverse event considered to be 'at least possibly related to treatment' will be recorded. Frequency tables will be constructed and the number of patients reporting an adverse event of grade 3 or higher at least possibly related to treatment will be reported.
Time Frame: Up to 5 years
Population: All patients that received protocol treatment were evaluable for this endpoint.
Measure: Number; unit: participants
Arm/Group | Phase II
Number analyzed (Participants) | 22
participants
  Grade 3+ Adverse Event | 8
  Grade 4+ Adverse Event | 1

4. Secondary Outcome: Duration of Response (Phase II)
Description: Duration of response is defined for all evaluable patients with changes in disease burden that met the RECIST criteria for CR or PR on 2 consecutive evaluations at least 6-8 weeks apart as the date at which the CR or PR to the date progression is documented. The distribution of response durations will be estimated using the Kaplan-Meier method.
Time Frame: Up to 5 years
Population: No patients were eligible for this endpoint.
Arm/Group | Phase II
Number analyzed (Participants) | 0

5. Secondary Outcome: Progression Free Survival (PFS) (Phase II)
Description: Progression free survival is defined as the time from registration to documentation of disease progression. If a patient dies without a documentation of disease progression, the patient will be considered to have had tumor progression at the time of their death unless there is sufficient documented evidence to conclude no progression occurred prior to death. If the patient is declared to be a major treatment violation, the patient will be censored on the date the treatment violation was declared to have occurred. In the case of a patient starting treatment and then never returning for any evaluations, the patient will be censored for progression on the last day of therapy was administered. The distribution of progression-free survival times will be estimated using the Kaplan-Meier method.The distribution of PFS times will be estimated using the Kaplan-Meier method.
Time Frame: Time from registration to documentation of disease progression, up to 5 years
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase II
Number analyzed (Participants) | 21
months | 2.0 [1.5 to 3.0]

6. Secondary Outcome: Progression Free Survival Rate
Description: Progression free survival (PFS) is defined as the time from registration to documentation of disease progression. A point and interval estimate of the 6 month PFS rate will be obtained using the Kaplan-Meier method.
Time Frame: At 6 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Phase II
Number analyzed (Participants) | 21
percentage of patients | 14.3 [5.0 to 40.7]

7. Secondary Outcome: Survival Time (Phase II)
Description: Survival time is defined as the time from registration to death due to any cause. The distribution of survival time will be estimated using the method of Kaplan-Meier.
Time Frame: Time from registration to death due to any cause
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase II
Number analyzed (Participants) | 21
months | 10.1 [4.9 to 19.1]

ADVERSE EVENTS:
Description: All patients that registered and started protocol treatment were available for adverse events assessment. Adverse Events were assessed during each cycle of treatment.
Groups:
- Dose Level 1; Dose Level -1; Dose Level -2; Dose Level -2A; Dose Level -2B: Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
- Phase II: laboratory biomarker analysis: Correlative studies
Arm/Group | Dose Level 1 | Dose Level -1 | Dose Level -2 | Dose Level -2A | Dose Level -2B | Phase II
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/2 | 1/7 | 3/6 | 3/8 | 7/22
Other Adverse Events (participants affected / at risk) | 3/3 | 2/2 | 7/7 | 6/6 | 8/8 | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 (N=3) | Dose Level -1 (N=2) | Dose Level -2 (N=7) | Dose Level -2A (N=6) | Dose Level -2B (N=8) | Phase II (N=22)
Hemoglobin decreased (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood glucose increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Protein urine positive (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 (N=3) | Dose Level -1 (N=2) | Dose Level -2 (N=7) | Dose Level -2A (N=6) | Dose Level -2B (N=8) | Phase II (N=22)
Hemoglobin decreased (Blood and lymphatic system disorders) | 3 (3) | 2 (3) | 5 (13) | 6 (15) | 5 (10) | 16 (42)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flashing vision (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 4 (6)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (5) | 3 (4) | 0 (0) | 9 (17)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Mucositis oral (Gastrointestinal disorders) | 3 (5) | 0 (0) | 6 (12) | 3 (7) | 5 (6) | 12 (21)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 3 (4) | 2 (3) | 10 (17)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 8 (11)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Fatigue (General disorders) | 3 (5) | 0 (0) | 6 (12) | 6 (16) | 6 (9) | 19 (52)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (3)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 4 (5)
Alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 6 (8)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (3) | 7 (10)
Bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 8 (14)
Leukocyte count decreased (Investigations) | 1 (1) | 1 (2) | 5 (8) | 5 (16) | 3 (4) | 13 (32)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (2) | 2 (2) | 3 (9) | 0 (0) | 4 (9)
Neutrophil count decreased (Investigations) | 1 (1) | 1 (2) | 5 (6) | 5 (10) | 2 (3) | 10 (24)
Platelet count decreased (Investigations) | 2 (2) | 2 (3) | 3 (9) | 3 (7) | 3 (7) | 13 (30)
Serum cholesterol increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 2 (4) | 0 (0) | 4 (5)
Weight loss (Investigations) | 1 (1) | 1 (1) | 4 (6) | 2 (9) | 1 (2) | 8 (20)
Anorexia (Metabolism and nutrition disorders) | 3 (5) | 1 (1) | 3 (5) | 5 (9) | 4 (5) | 14 (31)
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood glucose increased (Metabolism and nutrition disorders) | 3 (3) | 2 (2) | 4 (11) | 6 (18) | 4 (6) | 16 (39)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Serum albumin decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Serum calcium decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Serum calcium increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Serum potassium decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Serum sodium decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Serum triglycerides increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (4) | 2 (7) | 1 (1) | 8 (13)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (4)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (6)
Sinus pain (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Taste alteration (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Glomerular filtration rate decreased (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Protein urine positive (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ureteric obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Atrophy skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (8)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (5) | 0 (0) | 2 (4) | 1 (6) | 0 (0) | 5 (12)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash desquamating (Skin and subcutaneous tissue disorders) | 3 (5) | 1 (1) | 4 (7) | 3 (8) | 4 (5) | 11 (20)
Sweating (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (6)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less